CLINICAL TRIAL: NCT02945319
Title: Integrated Molecular and Clinical Profiling to Optimize Outcome Prediction in Splenic Marginal Zone Lymphoma
Status: Completed | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG46; NCT03288415 (obsolete NCT alias)
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Splenic Marginal Zone Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims at developing and validating an integrated clinico-molecular model for an accurate survival prognostication in newly diagnosed SMZL.

Already existing and coded tumor biological material and health-related personal data will be retrospectively collected. Mutation analysis will be performed by targeted deep next generation sequencing of tumor genomic DNA. Deletion of 7q will be assessed by FISH on nuclei isolated from tumor tissues. Immunoglobulin gene rearrangement and mutation status will be analyzed on tumor genomic DNA by PCR and Sanger sequencing. The methylation status of target genes will be assessed by methylation specific PCR on tumor genomic DNA.

The adjusted association between exposure variables and OS will be estimated by Cox regression. This approach will provide the covariates independently associated with OS that will be utilized in the development of a hierarchical molecular model to predict OS. The hierarchical order of relevance in predicting OS among covariates will be established by recursive partitioning analysis. An amalgamation algorithm will be used to merge terminal nodes showing homogenous OS. The discrimination capacity of the model will be assessed by calculating the c-index. Relative survival analysis will be used to provide a measure of the excess mortality experienced by patient's subgroups stratified according to the developed hierarchical molecular models, irrespective of whether the excess mortality is directly or indirectly attributable to the disease. The model developed in the training set will be tested in the validation sets and the model performance (c-index) in the validation set will be compared with that in the training set.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years or older
* Diagnosis of SMZL on spleen histology before Dec 31st 2010 (to provide the cohort with a minimum follow-up of at least 5 years)
* Availability of tumor material (from spleen, peripheral blood or bone marrow) collected before initiation of medical therapy
* Availability of the baseline and follow-up annotations

Exclusion Criteria:

* Having received any medical therapy including anti CD20 monoclonal antibody, chemotherapy or biological agents before splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of SMZL on spleen histology.
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of enrollment to study ending at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IOSI, Bellinzona, Switzerland